CLINICAL TRIAL: NCT07127991
Title: Impact of Neuromuscular Electrical Stimulation on Muscle Mass, Strength, and Functionality in Critically Ill Oldest Old Patients: a Randomized Controlled Trial
Brief Title: Neuromuscular Electrical Stimulation in Critically Ill Patients Aged 80 and Over
Acronym: NMES-ICU80
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Associate Professor in the Department of Rehabilitation Sciences, Faculty of Medicine, Universidad de La Frontera, Temuco, Chile., Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 234
Record Dates: First submitted 2025-08-01; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Units (ICUs); Muscle Atrophy or Weakness; Old and Very Old People
Keywords: MUSCLE ATROPHY; FUNCTIONAL STATUS; ICU; OLDER ADULTS; NMES
MeSH Terms: conditions — Muscular Atrophy; Asthenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking will be single-blind. The data analyst will receive the database with groups coded as A/B and will not have access to the allocation key until the primary analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (Other): Participants of the fourth age (≥80 years old) will receive the standard physical therapy routinely provided during their hospitalization. This intervention involves passive mobilization of the lower limbs, specifically within the ranges of hip flexion, knee flexion and extension, and ankle flexion and extension. One set of 10 bilateral repetitions will be performed while the patient is under sedation in the ICU. Once the patient is awake, the mobilization protocol routinely used in the same unit will be followed.
  This intervention will be carried out twice a day: the first session in the morning (08:00-12:00 hrs) and the second in the afternoon (14:00-18:00 hrs). This corresponds to the standard practice in the ICU of Dr. Hernán Henríquez Aravena Hospital.
  Interventions: Procedure: Standard physical therapy
- NMES GROUP (Experimental): The participant will receive standard physical therapy plus medium-frequency NMES.
  Two sessions will be carried out-one in the morning (08:00-12:00 hrs) and another in the afternoon (14:00-18:00 hrs)-always following standard physical therapy.
  Interventions: Device: Medium Frequency Neuromuscular Electrical Stimulation (NMES); Procedure: Standard physical therapy

INTERVENTIONS:
Device: Medium Frequency Neuromuscular Electrical Stimulation (NMES) — The medium-frequency NMES protocol, as reported in previous studies, consists of a carrier frequency of 2,500 Hz, a treatment frequency of 100 Hz, an ON time of 5 seconds (1 second ramp-up, 3 seconds contraction, and 1 second ramp-down), and an OFF time of 10 seconds. This stimulation protocol will be applied for 20 minutes per session (40 minutes of NMES per treatment day).
  Two electrodes will be placed on each thigh, located at the motor point of the quadriceps muscle. Electrode positions will be marked with a semi-permanent marker to ensure consistent placement across sessions.
  Arms: NMES GROUP
Procedure: Standard physical therapy — Participants of the fourth age (≥80 years old) will receive the standard physical therapy routinely provided during their hospitalization. This intervention involves passive mobilization of the lower limbs, specifically within the ranges of hip flexion, knee flexion and extension, and ankle flexion and extension. One set of 10 bilateral repetitions will be performed while the patient is under sedation in the ICU. Once the patient is awake, the mobilization protocol routinely used in the same unit will be followed.

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness of Medium-Frequency Neuromuscular Electrical Stimulation, in combination with standard physical therapy, compared to standard physical therapy alone, on muscle mass, muscle strength, and functionality in critically ill patients aged 80 and over during their hospital stay. The safety of the intervention and the standardization of protocol parameters will also be assessed.

The main research questions are:

* Does the implementation of a standardized Medium-Frequency Neuromuscular Electrical Stimulation protocol, in combination with standard physical therapy, compared to standard physical therapy alone, help attenuate the loss of skeletal muscle mass, strength, and functionality in critically ill patients aged 80 and over?
* Is the use of this protocol and its proposed parameters safe for critically ill patients aged 80 and over? The study will consist of applying a standardized Medium-Frequency Neuromuscular Electrical Stimulation protocol to oldest old patients admitted to the Intensive Care Unit of Dr. Hernán Henríquez Aravena Hospital in Temuco, Chile. The sample will consist of oldest old participants (≥80 years), who will be randomly divided into two subgroups: a control group that will receive standard physical therapy typically provided during hospitalization, and an experimental group that will receive the same standard therapy plus Medium-Frequency Neuromuscular Electrical Stimulation, which will begin within the first 48 hours of Intensive Care Unit admission.

The following variables will be assessed in both groups (control and experimental), from Intensive Care Unit admission to hospital discharge:

* Skeletal muscle mass characteristics and evolution (quadriceps femoris and anterior tibialis muscle thickness), measured by ultrasonography.
* Handgrip strength, measured using a digital hand dynamometer.
* Inspiratory muscle strength, assessed using a pimometer.
* Peripheral muscle strength, evaluated with the Medical Research Council Sum Score (MRC-SS).
* Functionality, assessed by the Functional Status Score for the Intensive Care Unit (FSS-ICU) .
* Independence in basic activities of daily living, measured using the Barthel Index.
* Quality of life, evaluated using the Short Form-36 Health Survey (SF-36).
* Cognitive impairment, assessed through the Montreal Cognitive Assessment (MoCA).
* Frailty, measured using the Clinical Frailty Scale (CFS).

DETAILED DESCRIPTION:
A clinical trial is proposed to evaluate the effectiveness of Medium-Frequency Neuromuscular Electrical Stimulation, in combination with standard physical therapy, compared to standard physical therapy alone on muscle mass, muscle strength, and functionality in critically ill patients aged 80 and over during their hospital stay. The study will also assess the safety of the intervention and the standardization of the parameters used in the protocol.

General Aim

To evaluate the effectiveness of medium-frequency neuromuscular electrical stimulation, in combination with standard physical therapy, versus standard physical therapy alone, on muscle mass, muscle strength, and functionality in critically ill oldest old patients during their hospital stay.

Specific Objectives

To compare quadriceps femoris muscle thickness (rectus femoris-vastus intermedius) and tibialis anterior muscle thickness via ultrasonography between the study groups during hospitalization.

To compare global peripheral muscle strength using the Medical Research Council Sum Score (MRC-SS) and handgrip strength using dynamometry between the study groups during hospitalization.

To compare maximal inspiratory muscle strength using pimometry between the study groups during hospitalization.

To compare patients' functional status using the Functional Status Score for the Intensive Care Unit (FSS-ICU) between the study groups during hospitalization.

To compare differences in levels of independence in activities of daily living using the Barthel Index between the study groups during hospitalization.

To compare health-related quality of life using the SF-36 questionnaire between the study groups during hospitalization.

To compare cognitive impairment using the Montreal Cognitive Assessment (MoCA) between the study groups during hospitalization.

To compare frailty levels using the Clinical Frailty Scale (CFS) between the study groups during hospitalization.

Methodology

A prospective, randomized controlled clinical trial is proposed, consisting of the application of a standardized medium-frequency neuromuscular electrical stimulation (NMES) protocol in oldest old patients admitted to the medical and surgical Intensive Care Units of Dr. Hernán Henríquez Aravena Hospital. The sample will consist of oldest old participants (≥80 years), who will be randomly divided into two subgroups: a control group (standard physical therapy) and an experimental group (standard therapy + NMES).

The control group will receive the standard physical therapy routinely provided during hospitalization. The experimental group will receive standard physical therapy plus medium-frequency NMES, which will begin within the first 48 hours of admission to the unit.

Population and Sample

The target and accessible population will include oldest old patients admitted to the Adult Critical Care Unit (ICU) at Dr. Hernán Henríquez Aravena Hospital in Temuco, Chile. Participant selection will be non-probabilistic, with patients being included as they meet the inclusion criteria. Once eligibility is confirmed, participants will be randomized into either the control group or the intervention group.

The recruitment process will begin once approval has been obtained from the hospital administration, the ethics committee, and the head of the Adult Intensive Critical Care Unit (ICU). The ICU staff will be notified of the start of data collection for patients meeting the inclusion criteria. The invitation to participate in the study will be extended by a collaborating physiotherapist who works permanently in the Adult ICU of Dr. Hernán Henríquez Aravena Hospital in Temuco, Chile. As eligible candidates are identified, they will be recruited into the study.

The recruitment site will be the Adult ICU facilities, including both the medical and surgical units, from admission until hospital discharge.

Sample Size Calculation

The sample size (N) was calculated using a statistical power of 80% and a significance level of 0.05, using the G*Power 3.1.9.7 software. The calculation was based on the variation in quadriceps muscle thickness (rectus femoris-vastus intermedius), measured via ultrasonography and expressed as a percentage, which was defined as the primary outcome variable.

According to previous studies, it is expected that muscle thickness will decrease significantly less in the group receiving medium-frequency NMES after the intervention period, with an estimated reduction of ~20% compared to the control group.

Based on the sample size calculation and for the purpose of assigning patients to the two described groups (control and medium-frequency NMES), a minimum of 24 patients (12 per group) is required to detect a difference in quadriceps muscle thickness changes (rectus femoris-vastus intermedius).

Considering an anticipated 20% dropout rate during the trial-due to the critical condition of the participants-the final number of participants expected to be recruited is 15 per group.

Intervention

The interventions will be carried out by the principal investigator and trained assistants during the research period. Prior to their application, pharmacological, ventilatory, and hemodynamic data will be recorded in order to assess the patient's condition and their response during mobilization and/or the application of electrical stimulation.

A. Standard Physical Therapy

All participants will receive standard physical therapy. This intervention includes passive mobilization of the lower limbs, specifically targeting the ranges of hip flexion, knee flexion and extension, and ankle flexion and extension. One set of 10 bilateral repetitions will be performed while the patient is under sedation in the ICU. Once the patient is awake, the mobilization protocol routinely used in the unit will be followed.

This intervention will be conducted twice daily: once in the morning shift (08:00-12:00 hrs) and once in the afternoon shift (14:00-18:00 hrs), consistent with routine ICU practices at Dr. Hernán Henríquez Aravena Hospital.

B. Medium-Frequency Neuromuscular Electrical Stimulation (NMES)

The NMES protocol involves the use of a 4-channel device (Enraf-Nonius®, Rotterdam, Netherlands), provided by the Muscle Mass and Strength Regulation Research Group at Universidad de La Frontera. Two sessions will be conducted daily-one in the morning (08:00-12:00 hrs) and one in the afternoon (14:00-18:00 hrs)-always after standard physical therapy.

Two electrodes will be applied to each thigh, placed at the motor point of the quadriceps muscle. This point has been identified in previous studies and is located by measuring the distance between the anterior superior iliac spine (ASIS) and the superior border of the patella. The midpoint of this measurement is identified, and from there, 5 cm proximally and 10 cm distally are marked. The electrodes will be positioned at these points, creating a 15 cm distance between them.

Electrode placement will be marked using a semi-permanent marker to ensure consistency across sessions.

The medium-frequency NMES protocol, as reported in previous studies, consists of a carrier frequency of 2,500 Hz, a treatment frequency of 100 Hz, an ON period of 5 seconds (1 second ramp-up, 3 seconds contraction, and 1 second ramp-down), and an OFF period (rest) of 10 seconds. Each session will last 20 minutes, totaling 40 minutes of NMES per treatment day.

Stimulation intensity will be set once a visible and palpable muscle contraction is achieved. The intensity will be adjusted every 3 minutes to maintain consistent stimulation throughout the session. The stimulation intensity (in mA) at the start and end of muscle contraction will be recorded in a data sheet.

Evaluations

The characteristics and progression of skeletal muscle mass (thickness of the quadriceps femoris and anterior tibialis muscles) will be assessed using ultrasonography. Handgrip strength will be measured using a digital hand dynamometer; inspiratory muscle strength will be evaluated using a pimometer; peripheral muscle strength will be assessed using the Medical Research Council Sum Score (MRC-SS); functionality will be assessed using the Functional Status Score for the Intensive Care Unit (FSS-ICU); independence in basic activities of daily living will be measured using the Barthel Index; quality of life will be assessed with the Short Form-36 Health Survey (SF-36); cognitive impairment will be evaluated using the MoCA (Montreal Cognitive Assessment); and frailty will be assessed with the Clinical Frailty Scale (CFS). These evaluations will be applied in both groups (control and experimental) from ICU admission to hospital discharge.

Quadriceps muscle thickness will be assessed at four specific time points:

ICU admission (baseline): within the first 24 hours after ICU admission (Day 1).

During ICU stay (intermediate ICU assessment): at the first occurrence when the patient reaches a level of consciousness sufficient for active participation, defined as a score ≥ 3 out of 5 on the "S5Q" scale, assessed daily (average: 5-6 days).

Prior to step-down unit discharge (end-of-ICU assessment): within the 12 hours preceding discharge from the ICU (average: 12-14 days).

Prior to hospital discharge (final assessment): within the 12 hours preceding hospital discharge (average: 18-20 days).

As for the evaluations of handgrip strength, pimometry, MRC-SS:

* During ICU stay (intermediate ICU assessment): at the first occurrence when the patient reaches a level of consciousness sufficient for active participation, defined as a score ≥ 3 out of 5 on the "S5Q" scale, assessed daily (average: 5-6 days).
* Prior to step-down unit discharge (end-of-ICU assessment): within the 12 hours preceding discharge from the ICU (average: 12-14 days).
* Prior to hospital discharge (final assessment): within the 12 hours preceding hospital discharge (average: 18-20 days).

FSS-ICU:

* During ICU stay (intermediate ICU assessment): at the first occurrence when the patient reaches a level of consciousness sufficient for active participation, defined as a score ≥ 3 out of 5 on the "S5Q" scale, assessed daily (average: 5-6 days).
* Prior to step-down unit discharge (end-of-ICU assessment): within the 12 hours preceding discharge from the ICU (average: 12-14 days).

The Barthel Index, SF-36 questionnaire, and MoCA test:

* Prior to step-down unit discharge (end-of-ICU assessment): within the 12 hours preceding discharge from the ICU (average: 12-14 days).
* Prior to hospital discharge (final assessment): within the 12 hours preceding hospital discharge (average: 18-20 days).

Frailty (CFS) will be assessed at the time of patient admission. Since patients are typically sedated at this stage, this scale allows for the objective identification of a frailty level through brief questions asked to the participant's caregiver.

Baseline characteristics of the participants will be obtained by reviewing their medical records.

Additionally, data collected at ICU admission will include the medical diagnosis, severity score using the Acute Physiology And Chronic Health Evaluation II (APACHE II), and the Clinical Frailty Scale score. Based on the information obtained upon admission, values such as Body Mass Index (BMI), comorbidities, surgical history, pharmacological treatments used, daily laboratory tests (e.g., CRP, CK, lipid profile), hemodynamic records during the intervention, fluid balance, length of ICU and hospital stay, days on mechanical ventilation, and motor milestones achieved will be recorded, among others.

As a data collection tool, a database will be created exclusively for this study. All data will be anonymized and coded; therefore, no identity will be disclosed. Physical documents (evolution charts and others) will be stored within the Adult Critical Care Unit of the Dr. Hernán Henríquez Aravena Hospital, and the digital data (database) will be stored on a computer designated exclusively for this project. Only the research team will have access to this device, ensuring the security of personal data and preventing unauthorized access, alteration, loss, or disclosure.

The personal and/or sensitive data of the study participants will not be disclosed, and the research team commits to upholding the confidentiality and privacy of all accessed information.

Participant Authorization

Patients will be invited to participate in the study (an action carried out by a collaborating physical therapist), and authorization will be requested to use the data recorded during their ICU stay, as well as data extracted from their medical records. This process will occur once the individual is alert, responsive, and cooperative, as determined by the Glasgow Coma Scale. A Glasgow score between 13 and 15 will be considered optimal, indicating the patient is capable of understanding and responding to verbal commands with an adequate level of consciousness. This Glasgow score will be obtained from the patient's daily evaluations, which are recorded in their medical chart. Once the patient has signed the informed consent, thus agreeing to participate in the study, data extraction from their clinical record will proceed.

Analysis Plan

The primary outcome will be defined as the occurrence of clinically significant deterioration in at least one of the three domains evaluated at ICU discharge:

1. skeletal muscle mass - ≥10% reduction in quadriceps thickness measured by ultrasound;
2. muscle strength - MRC-SS <48 points or ≥6 kg decrease in handgrip strength;
3. functionality - FSS-ICU <20 points or Barthel Index ≤60.

These continuous variables will be dichotomized based on validated cut-off points. For each individual component and for the composite outcome, the following will be calculated: relative risk (RR), absolute risk reduction (ARR), relative risk reduction (RRR), and number needed to treat (NNT), all with 95% confidence intervals. Rates will be estimated using binomial regression adjusted for age, sex, APACHE II score, and number of days on mechanical ventilation, thereby providing easily interpretable effect measures to quantify the clinical impact of NMES on muscle mass, strength, and function in critically ill older adults.

Data will be recorded in Microsoft Excel® and analyzed using IBM SPSS Statistics 30.0®. Results will be expressed as mean ± standard deviation for continuous variables and as frequency and percentage for categorical variables. The Shapiro-Wilk test will be used to assess data normality. The independent samples t-test will be used to compare means between groups (e.g., baseline characteristics). Repeated measures ANOVA will be used to assess the effects of time, group, and time × group interaction between the control and intervention groups. In the presence of a significant interaction, the paired samples t-test will be applied. Percentage change (delta) of outcome variables will also be calculated and compared using the independent samples t-test. In the intervention group, comparisons between muscles (quadriceps and tibialis anterior) will be conducted using the independent samples t-test. A p-value < 0.05 will be considered statistically significant.

Expected Results

This study aims to identify the impact of medium-frequency neuromuscular electrical stimulation on muscle mass loss, muscle strength, and functionality in critically ill patients in the fourth age during hospitalization.

It is anticipated that medium-frequency NMES will demonstrate measurable benefits in preserving muscle mass and strength, and in accelerating functional recovery, without compromising the safety of patients aged 80 and older.

Based on the results, the study intends to propose early intervention strategies for patients in the fourth age.

ELIGIBILITY:
Inclusion Criteria:

* People aged 80 years or older.
* Hospitalized in the Adult Critical Care Unit of Dr. Hernán Henríquez Aravena Hospital in Temuco.
* Estimated mechanical ventilation time greater than 72 hours.

Exclusion Criteria:

* Patients with prior neurological complications.
* Patients with severe dependence prior to admission.
* Patients with difficult-to-manage hemodynamic instability.
* Patients with accessory elements that limit assessment.
* Patients with lower limb amputation.
* Patients in the prone position.
* Patients with loss of skin integrity.
* Patients expected to remain in the unit for less than 72 hours.

Patients transferred from other services with a stay of more than 72 hours.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Skeletal Muscle Mass | ICU admission (baseline): Day 1 During ICU stay (intermediate ICU assessment): average: Day 4-6 Prior to step-down unit discharge (end-of-ICU assessment): average: Day 12-14 Prior to hospital discharge (final assessment): average: Day 18-20
  For the assessment of muscle mass, the thickness of the quadriceps muscle-composed of the vastus intermedius and rectus femoris-and the anterior tibialis muscle will be measured using ultrasonography.
  For quadriceps thickness, the reference point will be the midpoint between the anterior superior iliac spine and the superior pole of the patella. At this point, the following measurements will be taken: vastus intermedius (VI), rectus femoris (RF), and total quadriceps thickness (TQ).
  For the anterior tibialis muscle, the reference point will be the first third of the distance between the lateral condyle of the tibia and the upper edge of the lateral malleolus. At this reference point, the image will be frozen and the thickness of the anterior tibialis muscle will be measured. For each muscle, three consecutive measurements will be taken, and the average value will be recorded in centimeters.

SECONDARY OUTCOMES:
Change in Handgrip Strength | During ICU stay (intermediate ICU assessment): on average Day 4-6 Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average Day 18-20
  Handgrip strength (HS) will be assessed using a JAMAR® digital dynamometer. Grip strength will be measured in both the dominant and non-dominant hands. During the assessment, the participant will be in a long sitting position (sitting upright in bed), with shoulders adducted and without rotation, the elbow flexed at 90° close to the body, and the forearm and wrist in a neutral position. The assessed arm will be supported on a pillow. The examiner will hold the dynamometer in a vertical position, and the participant will exert their maximum grip strength for 3 seconds. Grip strength will be measured three times on each hand alternately, and the highest recorded value will be used for analysis.
Change in Peripheral Muscle Strength | During ICU stay (intermediate ICU assessment): on average Day 4-6 Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average Day 18-20
  Peripheral muscle strength will be assessed using the Medical Research Council Sum Score (MRC-SS), which evaluates the global peripheral muscle strength of six major muscle groups during functional movements (shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, and ankle dorsiflexion) on each side of the body. Each group is rated from 0 (no visible contraction) to 5 (normal strength throughout the full range of motion). Each participant will be assigned a total score ranging from 0 (total paralysis) to 60 (normal strength).
  Assessments will be performed from right to left and from proximal to distal, following that same sequence. Up to three optimal attempts will be allowed per muscle group, with a rest period of at least 30 seconds between attempts.
Change in Inspiratory Muscle Strength | During ICU stay (intermediate ICU assessment): on average Day 4-6 Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average Day 18-20
  Inspiratory muscle strength will be assessed using a digital manometer (MicroRPM®, Vyaire Medical, Hoechberg, Germany). The evaluations will follow the American Thoracic Society (ATS) recommendations for respiratory muscle strength testing. Participants will be instructed to:
  i) perform a rapid exhalation down to residual volume, and ii) execute a maximal inhalation "with as much force as possible." The result from this measurement will be compared against predictive equations for maximal respiratory pressures, which vary based on sex and age. The highest value from three maneuvers with less than 10% variation will be recorded, with a 1-minute rest between each attempt.
Change in ICU Functionality | During ICU stay (intermediate ICU assessment): on average Day 4-6 Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14
  Functionality in the ICU will be assessed using the Chilean version of the Functional Status Score for the Intensive Care Unit (FSS-ICU). The FSS-ICU measures the level of physical assistance required for five functional activities in the intensive care setting: rolling in bed, transitioning from supine to sitting, sitting at the edge of the bed, transferring from the bed to standing, and walking. Walking will only be assessed if the participant is able to complete a 30-meter walk. Each activity is scored from 0 points (unable to perform) to 7 points (complete independence). The total score is the sum of the scores for each completed activity, with a higher score indicating greater functional mobility.
Change in Independence in Performing Activities of Daily Living | Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average Day 18-20
  The Barthel Index assesses the degree of independence in performing activities of daily living based on the level of assistance participants require to carry out the described tasks. The Barthel Index evaluates 10 basic activities of daily living (ADLs), assigning a score ranging from 0 (total dependence) to 100 (complete independence).
  The assessment will be conducted when the patient is awake and cooperative, with a score ≥ 3 on the S5Q test, which is evaluated daily.
Change in Perceived Health Status | Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average Day 18-20
  Quality of life will be assessed using the SF-36 (Short Form-36 Health Survey) questionnaire, which evaluates quality of life through questions related to functional status, emotional well-being, social functioning, and general health perception. The SF-36 contains 36 questions grouped into 8 domains: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. This scale has been described as a useful tool for evaluating outcomes after critical illness. The assessment will be performed when the patient is awake and cooperative, with a score of ≥ 3 on the S5Q test, evaluated daily.
Change in Frailty | ICU admission (baseline): Day 1 Prior to hospital discharge (final assessment): average: Day 18-20
  Frailty will be assessed using the Clinical Frailty Scale (CFS), a global 9-point scale based on clinical evaluation of mobility, energy, physical activity, and function. It provides a quick and simple way to assess a person's level of frailty and summarizes the physical fitness of older adults. The scale ranges from 1 point ("very fit") to 9 ("terminally ill"), with higher scores indicating greater risk. When applied in the context of acute illness or hospital admission-such as ICU admission-it is the only scale that allows interviewing the caregiver to objectively assess the patient's frailty level based on their premorbid status two weeks prior to the acute event.
Change in Cognitive Impairment | Prior to step-down unit discharge (end-of-ICU assessment): on average Day 12-14 Prior to hospital discharge (final assessment): on average 18-20
  Cognitive impairment will be assessed using the MoCA scale (Montreal Cognitive Assessment). This brief test is designed to detect mild cognitive impairment by evaluating multiple cognitive domains. It consists of 30 items that examine functions such as attention, memory, language, executive functions, visuospatial skills, abstraction, calculation, and orientation. The maximum total score is 30 points, and a score below 26 suggests cognitive impairment. In hospital settings or among individuals with low educational levels, 1 point may be added if the patient has ≤12 years of schooling. The assessment will be conducted when the patient is awake and cooperative, with a score ≥ 3 on the S5Q test, which is evaluated daily.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Nasri Marzuca-Nassr, PhD, Study Chair — Universidad de La Frontera
Locations (1):
- Hospital Dr Hernán Henríquez Aravena, Temuco, Región de la Araucanía, Chile

IPD SHARING:
Plan to Share IPD: No
IPD Sharing Plan Description:
  All individual participant data (IPD) that underlie the results reported in future publications, including anonymized demographic, clinical, and outcome variables, will be made available. Data dictionaries describing each variable will also be provided. The data will be shared with qualified researchers upon reasonable request after study completion and publication, through a controlled-access repository or direct agreement with the principal investigator, in compliance with applicable ethical and legal requirements.

REFERENCES:
- [Background] Wageck B, Nunes GS, Silva FL, Damasceno MC, de Noronha M. Application and effects of neuromuscular electrical stimulation in critically ill patients: systematic review. Med Intensiva. 2014 Oct;38(7):444-54. doi: 10.1016/j.medin.2013.12.003. Epub 2014 Jul 22. PMID 25060511